CLINICAL TRIAL: NCT00984243
Title: An Evaluation of the Effectiveness of Photodynamic Therapy (PDT) Compared to Surgical Resection in Early Stage Roentgenographically Occult Lung Cancer.
Brief Title: Photodynamic Therapy (PDT) in Lung Cancer
Acronym: PDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Eric S. Edell, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 281-92; PulmMed 649
Record Dates: First submitted 2007-12-24; First posted 2009-09-25 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Photodynamic Therapy (Experimental): PHOTODYNAMIC THERAPY (PDT)
  Interventions: Procedure: PHOTODYNAMIC THERAPY (PDT)

INTERVENTIONS:
Procedure: PHOTODYNAMIC THERAPY (PDT) — Photodynamic Procedure:
  Photofrin II will be injected at a dosage of 2 mm/Kg intravenously. Laser treatment will take place 40-50 hours later. An argon-dye or an excimer-dye laser tuned to 620-630 nm will be used.
  It is anticipated that a microlens fiber will be used in almost all cases, but a cylinder-diffusing fiber can be used to treat lesions in segmental bronchi if needed.
  Argon-dye laser: Power settings 200 milliwatt (mW) microlens and 400 mW for cylinder Excimer laser: 4 milliJoules (mJoules)/pulse at 30 hertz for the microlens
  Energy density:
  Argon-dye laser: 200-300 Joules/cm^2 Excimer-dye laser: 100-200 Joules/cm^2

SUMMARY:
This study is being done to determine whether a substance called hematoporphyrin can be used to treat tumors in various locations in the body when used in association with a laser. Hematoporphyrin is a substance that is taken up by cancerous cells. When these cells are exposed to the energy emitted by a laser source, chemical reactions occur in the cell and cause the cells to die. It is hoped that this treatment method may be able to selectively destroy malignant cells without damaging surrounding healthy tissue.

DETAILED DESCRIPTION:
Lung cancer is currently the leading cause of death in both women and men in the United States and continues to be a major problem in several other countries in the world. Detection, localization, and surgical treatment at an early stage, provides the best opportunity for long-term survival for patients with non-sma11 cell lung cancer at this time. Studies examining the utility of screening patients at high risk for lung cancer with sputum cytology and chest roentgenograms showed that, despite a higher frequency of detecting and resecting early cancers in the screened group, there was no difference between the screened group and the control group in overall cancer mortality.

The purpose of this study is to determine if photodynamic therapy (PDT) is an alternative to surgical resection in patients with early stage) roentgenographically occult squamous cell carcinoma of the lung who are candidates for surgery. If PDT is successful, it would remove the indication for surgery and eliminate the need for an operation. The specific goals are to evaluate the impact of PDT on these patients by determining the percentage of patients who are spared surgery as wel1 as the following: morbidity, overall mortality, lung cancer mortality, the rate of subsequent lung cancer, the relative cost of PDT and surgery, the change in pulmonary function over time, the effect on quality of life, and the patient preferences for PDT and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient less than 75 years of age.
* Squamous cell lung cancer proven by biopsy or repeated Brushings obtained from the same location at separate bronchoscopies.
* Occult lung cancer by chest roentgenogram and CT scan If CT scan is abnormal, mediastinoscopy is negative.
* Cancer is bronchoscopically superficial as defined in section IV, E.
* Estimated size less than 1 cm diameter on the surface of the bronchus with the surface area of 0.7 to 1.0 cm2.
* Location in the trachea, main stem bronChi, lobar bronchi, segmental bronchi, or subsegmental bronchi.
* Medical condition permits surgery: cardiovascular status is satisfactory for operation and postoperative FEVl is predicted to be greater than 0.75 liter.
* Patients will complete quality of life questionnaire and a spirometry which will include forced expiratory volume in 1 second (FEVl) and forced vital capacity (FVC).
* On bronchoscopic biopsy, the carcinoma is entirely in situ or shows no more than 2 mm of microinvasion.
* The characteristics of the mucosa. may include paleness, opacity, loss of luster, roughness, micro-granularity.
* The mucosal folds may demonstrate lack of clarity. thickening, disappearance.
* There may be small nodular protrusion of tumor into the lumen
* The peripheral extent of tumor invasion can be confirmed endoscopically.

Exclusion Criteria:

* A medical disease which excludes surgery as an option
* A postoperative FEVl predicted to be less than 0.75 liter
* A previous carcinoma or other malignancy not curatively treated
* The presence of simultaneous lung cancers
* CT scan of the chest shows thickening of the bronchial wall or extension beyond the bronchial wall in the area of the cancer

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1994-02; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of PDT on these patients by determining the percentage of patients who are spared surgery. | 3 years

SECONDARY OUTCOMES:
Morbidity,overall mortality and lung cancer mortality. | 3 years
Rate of subsequent lung cancer. | 3 years
Relative cost of PDT and surgery. | 3 years
Change in pulmonary function over time. | 3 years
Effect on quality of life. | 3 years
Patient preferences for PDT and surgery. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric S. Edell, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States